CLINICAL TRIAL: NCT00477035
Title: A Phase I Study of Post-transplant Autologous Cytokine-induced Killer (CIK) Cells for the Treatment of High-risk Hematologic Malignancies
Brief Title: Post-transplant Autologous Cytokine-induced Killer (CIK) Cells for Treatment of High Risk Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sally Arai (Other)
Responsible Party: Sponsor-Investigator, Sally Arai, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-00245; 95889 (Other: Stanford University Alternate IRB Approval Number); BMT173 (Other: OnCore)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Leukemia; Multiple Myeloma
MeSH Terms: conditions — Leukemia; Multiple Myeloma | interventions — Etoposide; etoposide phosphate; Carmustine; Cyclophosphamide; Gemcitabine; Vinorelbine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Cytokine-induced Killer Cells (Experimental)
  Interventions: Drug: CIK cells; Drug: etoposide; Drug: bcnu; Drug: cyclophosphamide; Drug: gemcitabine; Drug: vinorelbine; Drug: melphalan

INTERVENTIONS:
Drug: CIK cells — 2x10e8 cells/kg
  Other Names: autologous cytokine-induced killer cells
Drug: etoposide — 60 mg/kg
  Other Names: Eposin; Etopophos; Vepesid; VP-16
Drug: bcnu — 15 mg/kg
  Other Names: Carmustine
Drug: cyclophosphamide — 100 mg/kg
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: gemcitabine — 1250 mg/m2
  Other Names: Gemzar
Drug: vinorelbine — 30 mg/m2
  Other Names: Navelbine
Drug: melphalan — 200 mg/m2
  Other Names: Alkeran; Melphalan hydrochloride

SUMMARY:
The purpose of the study is to conduct a phase I study of adoptive immunotherapy with autologous, ex-vivo expanded cytokine-induced killer (CIK) cells to reduce the relapse rate in autologous stem cell transplant patients with high-risk hematologic malignancies.

DETAILED DESCRIPTION:
Disease relapse remains the major cause of treatment failure in autologous stem cell transplantation for patients with high-risk disease. Relapse after autologous transplant is in part due to the persistence of residual cancer cells. Cellular immunotherapy using activated autologous effector cells to recognize and kill tumor targets in a minimal disease state after transplant is a strategy being explored to reduce relapse and improve survival. We hypothesize that cytokine-induced killer (CIK) cell-based immunotherapy can reduce the relapse rate after high-risk autologous stem cell transplantation by treating post-transplant minimal residual disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age, inclusive candidates for standard autologous SCT who are at high risk for relapse:

  * Acute myelogenous leukemia (AML), high risk, in CR1 or beyond without a donor (CR1 defined as: normal bone marrow morphology, resolution of any previously abnormal karyotype, neutrophils > 1000/ul, platelets > 100,000/ul, independence from red cell transfusion, no evidence extramedullary leukemia)
  * Hodgkin's lymphoma relapsed or refractory, with the presence of >= 1 adverse risk factor (Adverse risk factors are defined as stage IV involvement of the lung or bone marrow, constitutional symptoms, and the presence of more than minimal residual disease before the preparatory regimen)
  * Multiple myeloma with high risk features with only single autologous transplant option. High risk features defined as IgA myeloma, B2M > 2.5 mg/ml with normal kidney function, complex karyotypes or isolated chromosome 13 abnormalities, standard-dose therapy > 12 months, or inability to achieve at least 50% reduction of plasma cells in the bone marrow or 50% reduction in the paraprotein concentration after initial induction chemotherapy prior to transplant.
* Patients must have ECOG performance status < 2
* Patients must have adequate renal function with a serum creatinine of < 2 mg/dl or creatinine clearance > 50 ml/min.
* Patients must have adequate liver function with a total bilirubin < 2 mg/dl or transaminases < 3 times the upper limit of normal.
* Patients must have negative antibody serology for human immunodeficiency virus (HIV1 and 2)
* Adult women and minorities will be included. Patients with childbearing potential must use effective contraception.
* Patients must sign informed consent prior to initiation of any study-related treatments.

Exclusion Criteria:

* ECOG performance status > 2
* LVEF < 45%
* Pulmonary diffusion capacity < 50% predicted
* Total bilirubin > 2 mg/dl
* Creatinine > 2 mg/dl
* Pregnancy
* Patients positive for HIV
* Patients with engraftment failure at day 42 post transplant defined as failure to achieve a granulocyte count > 500/ul on 3 successive daily determinations and an unsupported platelet count of >= 50,000/ul by day 42
* Patients with active, uncontrolled infection that is expected to continue beyond day 42-63.
* Patients who fail to collect sufficient quantities of stem cells (> 1.6 x 10^9 cells) during apheresis to support CIK cell expansion cultures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To document the toxicities of infusion of autologous CIK cells | Day 42 post autologous stem cell transplant
Measure freedom from progression (FFP) | 1 and 2 years post-transplant
Measure event free survival | 1 and 2 years post-transplant
Measure overall survival | 1 and 2 years post-transplant

SECONDARY OUTCOMES:
Measure disease response | at day 40-60, day 90, day 180, and yearly

CONTACTS AND LOCATIONS:
Overall Officials: Sally Arai, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No